CLINICAL TRIAL: NCT05486208
Title: A Phase 1, Multicenter, Randomized, Placebo-Controlled, Double-Blind, Single-Ascending Dose Study of LY3844583 in Healthy Participants, and Multiple-Dose Study of LY3844583 in Healthy Participants and Patients With Atopic Dermatitis
Brief Title: A Study of LY3844583 in Healthy Participants and Participants With Atopic Dermatitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to lack of efficacy signal in atopic dermatitis participants.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18365; J3V-MC-KKAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-08-02; First posted 2022-08-03 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Healthy; Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LY3844583 (Part A) (Experimental): Single doses of LY3844583 administered subcutaneously (SC) and/or intravenously (IV).
  Interventions: Drug: LY3844583
- LY3844583 (Part B) (Experimental): Multiple doses of LY3844583 administered SC and/or IV.
  Interventions: Drug: LY3844583
- LY3844583 (Part C) (Experimental): Repeat doses of LY3844583 administered SC and/or IV.
  Interventions: Drug: LY3844583
- Placebo (Part A) (Placebo Comparator): Placebo administered SC and/or IV.
  Interventions: Drug: Placebo
- Placebo (Part B) (Placebo Comparator): Placebo administered SC and/or IV.
  Interventions: Drug: Placebo
- Placebo (Part C) (Placebo Comparator): Placebo administered SC and/or IV.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3844583 — Administered SC and/or IV.
  Arms: LY3844583 (Part A); LY3844583 (Part B); LY3844583 (Part C)
Drug: Placebo — Administered SC and/or IV.
  Arms: Placebo (Part A); Placebo (Part B); Placebo (Part C)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3844583 in healthy participants and participants with atopic dermatitis. The study will also assess how fast LY3844583 gets into the blood stream and how long it takes the body to remove it. The study is open to healthy participants and participants with atopic dermatitis. The study will be conducted in three parts and each participant will enroll in one part. The study will last up to 88, 116, and 186 days with 10, 13, and 14 visits for each participant in parts A, B, and C, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants (Parts A and B):

  * Are male or female not of childbearing potential
  * inclusion of healthy Japanese participants, the participant must be first-generation Japanese, defined as the participant's biological parents and all of the participant's biological grandparents must be of exclusive Japanese descent, and must have been born in Japan.
  * inclusion of healthy Chinse participants, the participant must be at a minimum, third-generation Chinese, defined as all 4 of the participants' biological grandparents must be of exclusive Chinese descent and born in China.
  * Must have a body mass index of 18.0 to 32.0 kilograms per meter squared (kg/m²), inclusive. For healthy Japanese participants, have a body mass index of 18.0 to 28.0 kg/m², inclusive, and a body weight of 50 kg to 85 kg, inclusive.
* Atopic dermatitis participants (Part C):

  * Must have a body mass index of 18.0 to 45.0 kg/m², inclusive
  * Are male or female participants including those of child bearing potential
  * Must have a diagnosis of AD for at least 12 months with either poor response to topical treatments or inability to use topical treatments
  * Must agree to use moisturizer daily throughout the treatment period

Exclusion Criteria:

* All participants:

  * Have or used to have health problems or laboratory test results or electrocardiogram (ECG) readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
  * Have active or latent tuberculosis
  * Have had any cancer within the past 5 years. Exceptions: successfully treated basal cell skin carcinoma or squamous cell skin carcinoma, with no evidence of recurrence or metastatic disease within the 3 years prior to baseline
  * Have one of the following viral infections: hepatitis B virus, hepatitis C virus or human immunodeficiency virus.
  * Have received treatment with biologic agents (such as monoclonal antibodies, including marketed drugs) within 30 days or 5 half-lives (whichever is longer) prior to dosing
  * Must not have previously completed a clinical trial with a molecule targeting interleukin-33 and/or the interleukin-33 receptor (ST2)
  * Are currently participating in or completed a clinical trial within the last 30 days
  * Have received a vaccine containing a live (attenuated) virus within 28 days of screening or intend to receive during the course of the study
* Atopic dermatitis participants:

  * Must not have received certain topical medications for AD within 2 weeks prior to randomization
  * Must not have received certain oral medications for AD or received phototherapy within 4 weeks prior to randomization
  * Must not have received any antibody-based biologic agents (marketed or investigational) within 5 half lives (t1/2) of the drug prior to randomization
  * Must not have received intravenous, intramuscular, or intra-articular steroids in the past 6 weeks prior to randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Adverse Events (AEs), Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Day 186
  A summary of AEs, TEAEs and SAEs, regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Concentration (Cmax) of LY3844583 | Pre-dose on Day 1 up to 186 days post-dose
  PK: Cmax of LY3844583
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3844583 | Pre-dose on Day 1 up to 186 days post-dose
  PK: AUC of LY3844583

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Parexel Early Phase Unit at Glendale, Glendale, California, United States
- Japan (2):
  - Medical Corporation Heishinkai OPHAC Hospital, Osaka, Osaka
  - P-one clinic, Hachiōji, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3844583 in Healthy Participants and Participants With Atopic Dermatitis — https://trials.lilly.com/en-US/trial/352936